CLINICAL TRIAL: NCT07285057
Title: Diagnostic Utility of rhPSMA-7.3 (18F) PET /CT Imaging in Patients With Prostate Cancer on Active Surveillance
Brief Title: Diagnostic Utility of rhPSMA-7.3 (18F) PET/CT in Men With Prostate Cancer on Active Surveillance
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Blue Earth Diagnostics (Industry)
Responsible Party: Principal Investigator, Ashutosh Kumar Tewari, Professor and System Chair, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY-25-00518
Record Dates: First submitted 2025-12-09; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Prostatic Neoplasms; Prostate Cancer; Prostate Adenocarcinoma
Keywords: Prostate cancer; Prostatic neoplasms; Active surveillance; PSMA PET/CT; rhPSMA-7.3; Prostate biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single-arm, prospective diagnostic imaging study in which all enrolled participants will undergo rhPSMA-7.3 (¹⁸F) PET/CT and standard multiparametric MRI prior to confirmatory prostate biopsy. Each participant serves as an own control for within-patient comparison of imaging modalities. No randomization or separate intervention arms are used.
Masking Description: This is an open-label diagnostic imaging study. Neither participants nor investigators are blinded to the imaging procedures. However, imaging interpretation will be performed independently - PET/CT scans will be reviewed by nuclear medicine physicians blinded to MRI findings, and MRI scans will be reviewed by radiologists blinded to PET/CT results. Pathologists evaluating biopsy specimens will be blinded to imaging results to minimize interpretation bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- rhPSMA-7.3 (18F) PET/CT Imaging (Experimental): Participants in this arm will undergo rhPSMA-7.3 (¹⁸F) PET/CT (flotufolastat F18, POSLUMA®) imaging and standard multiparametric MRI prior to confirmatory prostate biopsy. All participants receive the same imaging procedures; there are no control or comparison arms.
  Interventions: Radiation: rhPSMA-7.3 (18F) PET/CT Imaging (Flotufolastat F18, POSLUMA®); Drug: Flotufolastat F18

INTERVENTIONS:
Radiation: rhPSMA-7.3 (18F) PET/CT Imaging (Flotufolastat F18, POSLUMA®) — Participants will undergo a single rhPSMA-7.3 (¹⁸F) PET/CT scan using flotufolastat F18 (POSLUMA®), an FDA-approved PSMA-targeted radiotracer. The radiotracer will be administered intravenously at the standard diagnostic dose prior to PET/CT image acquisition. The scan will be performed according to institutional imaging protocols, approximately 50-70 minutes post-injection.
Drug: Flotufolastat F18 — An FDA-approved PSMA-targeted radiotracer. The radiotracer will be administered intravenously at the standard diagnostic dose prior to PET/CT image acquisition.
  Other Names: POSLUMA®

SUMMARY:
This investigator-initiated, prospective study evaluates the diagnostic utility of rhPSMA-7.3 (¹⁸F) PET/CT (flotufolastat F18, marketed as POSLUMA®) in men with biopsy-proven, low-risk or favorable intermediate-risk prostate cancer managed with active surveillance. The study aims to determine whether the addition of PSMA-based PET/CT to standard multiparametric MRI (mpMRI) improves detection of clinically significant prostate cancer compared to MRI alone. Eligible participants will undergo rhPSMA-7.3 (¹⁸F) PET/CT and mpMRI prior to confirmatory prostate biopsy. Biopsies will target areas identified on MRI, PET/CT, or both, and histopathologic outcomes will serve as the reference standard. The study will assess lesion-level concordance between PET/CT, MRI, and pathology, and evaluate the predictive value of PET/CT for disease upgrading. Approximately 120 participants will be enrolled at Mount Sinai Hospital over 12 months. Study participation will involve one imaging visit, one confirmatory biopsy, and follow-up through review of clinical results. There is minimal risk to participants beyond standard diagnostic procedures. The study is funded jointly by the Icahn School of Medicine at Mount Sinai and Blue Earth Diagnostics, which provides the imaging agent flotufolastat F18 and technical support.

DETAILED DESCRIPTION:
This investigator-initiated, single-center, prospective study aims to evaluate the diagnostic utility of rhPSMA-7.3 (¹⁸F) PET/CT (flotufolastat F18, marketed as POSLUMA®) in detecting clinically significant prostate cancer (csPCa) among men on active surveillance for low-risk or favorable intermediate-risk prostate cancer.

Background and Rationale: Active surveillance (AS) is the preferred management strategy for carefully selected men with low-risk and favorable intermediate-risk prostate cancer, balancing the avoidance of overtreatment against the need to identify disease progression early. Current surveillance strategies rely on serial PSA monitoring, digital rectal examination, mpMRI, and confirmatory biopsies. However, mpMRI can miss or underestimate clinically significant lesions, particularly those in the anterior or transitional zones. Prostate-specific membrane antigen (PSMA) is highly expressed in prostate cancer cells and can be visualized using PET/CT imaging with radiolabeled PSMA ligands. The next-generation tracer rhPSMA-7.3 (¹⁸F), or flotufolastat F18, has demonstrated improved image resolution, favorable kinetics, and low urinary excretion compared to earlier PSMA ligands. Incorporating PSMA PET/CT into the active surveillance pathway may identify occult or higher-grade disease not detected by MRI, improving risk stratification and treatment decision-making.

Study Objectives: The primary objective of the study is to determine whether the addition of rhPSMA-7.3 (¹⁸F) PET/CT to standard mpMRI improves detection of clinically significant prostate cancer (ISUP Grade Group ≥2) in men on active surveillance.

Secondary objectives include: Comparing lesion-level concordance between PET/CT, mpMRI, and histopathology. Evaluating the predictive value of PET SUVmax for detecting clinically significant disease. Assessing diagnostic performance metrics (sensitivity, specificity, PPV, NPV) for PET/CT versus MRI. Quantifying the proportion of patients reclassified (i.e., upgraded or transitioned from AS to definitive treatment) based on PET/CT findings.

Exploratory endpoints include: Association between PET quantitative parameters (SUVmax, lesion volume) and PSA density. Characterization of PET-only lesions not visualized on MRI. Correlation of PET/CT findings with adverse pathological features (ECE, SVI, cribriform/intraductal carcinoma) at biopsy or surgery. Evaluation of lesion-level changes in SUVmax and volume in patients who undergo repeat PET/CT.

Study Design: This is a prospective, single-arm diagnostic utility study. Approximately 120 participants with histologically confirmed low-risk or favorable intermediate-risk prostate cancer managed with active surveillance will be enrolled at Mount Sinai Hospital. All participants will undergo both mpMRI and rhPSMA-7.3 (¹⁸F) PET/CT prior to confirmatory biopsy. Imaging data will be reviewed by genitourinary radiologists and nuclear medicine physicians blinded to each other's findings. Lesions will be recorded according to standardized templates (e.g., PIRADS 2.1 for MRI and SUV-based mapping for PET/CT). Targeted biopsies will include MRI-positive, PET-positive, and fusion (concordant) targets, as well as systematic cores as per institutional protocol. Histopathology will serve as the reference standard for correlation. The study involves one PET/CT visit, one confirmatory biopsy, and up to three follow-up visits within 12 months.

Risks and Benefits: Risks include exposure to low-dose radiation comparable to standard diagnostic imaging, and expected biopsy-related discomfort such as pain, bleeding, infection, or transient urinary symptoms. Rare allergic reactions to flotufolastat F18 and mild emotional stress associated with imaging or awaiting results are possible but uncommon. There may be no direct benefit to participants. However, rhPSMA-7.3 (¹⁸F) PET/CT may help identify previously undetected higher-grade disease, leading to earlier or more appropriate treatment. The findings could improve future management of men on active surveillance.

Statistical Considerations: Diagnostic accuracy metrics will be analyzed at both lesion and patient levels using confirmatory biopsy as the gold standard. ROC analysis will determine SUVmax thresholds for predicting clinically significant disease. Concordance between PET and MRI findings will be evaluated with Cohen's kappa and McNemar's test. Sample size (n=120) is based on expected detection differences between PET/CT and MRI with 80% power and alpha=0.05.

Study Oversight: This study is conducted under the oversight of the Mount Sinai Program for the Protection of Human Subjects (PPHS) and complies with FDA regulations for IND-exempt studies involving FDA-approved radiopharmaceuticals (21 CFR 312.2(b)(1)). The study is jointly funded by the Icahn School of Medicine at Mount Sinai and Blue Earth Diagnostics. Mount Sinai is the study sponsor and holds regulatory responsibility. Blue Earth Diagnostics provides the imaging agent flotufolastat F18 (POSLUMA®), technical support, and partial financial support. Data management and analysis will be conducted internally at Mount Sinai. No external contract research organization (CRO) or vendor (e.g., Parexel) will manage study data.

Expected Duration: Enrollment start: November 2025 Primary completion: May 2027 (final confirmatory biopsy) Study completion: November 2027 (data lock and analysis)

Potential Impact: This study may validate the clinical role of rhPSMA-7.3 (¹⁸F) PET/CT in improving detection of clinically significant prostate cancer during active surveillance. The results may support integration of PSMA-targeted PET imaging into future diagnostic pathways, minimizing unnecessary biopsies and improving individualized management.

ELIGIBILITY:
Inclusion Criteria:

* Male participants aged ≥18 years.
* Histologically confirmed diagnosis of prostate adenocarcinoma.
* Classified as low-risk or favorable intermediate-risk prostate cancer according to NCCN criteria: Low-risk: Grade Group 1, PSA <10 ng/mL, cT1-T2a Favorable intermediate-risk: Grade Group 2, PSA 10-20 ng/mL, cT2b-c Currently managed with active surveillance.
* Able and willing to undergo rhPSMA-7.3 (¹⁸F) PET/CT imaging, mpMRI, and confirmatory prostate biopsy.
* Able to provide written informed consent.

Exclusion Criteria:

* A history of other active malignancy within the last 5 years, except for non-melanoma skin cancer.
* Contraindication to 3-T mpMRI.
* Significant intercurrent morbidity** limiting compliance with study protocols.

  ** Significant intercurrent morbidity refers to a substantial medical condition or complication that arises during a study or treatment, which is severe enough to impact the patient's participation, treatment outcomes, or overall prognosis. These conditions may be unrelated to the primary disease but can influence clinical decision-making, treatment efficacy, and patient safety. Examples include major infections, cardiovascular events, organ failure, or significant worsening of pre-existing comorbidities (https://doi.org/10.1016/S1053-4296(03)00031-6).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Agent(s) or other agents used in study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with Grade Group ≥ 2 | Up to 3 months after PET/CT imaging
  Detection rate measured by the proportion of participants with clinically significant prostate cancer (csPCa) (Grade Group ≥2) using rhPSMA-7.3 (¹⁸F) PET/CT compared to standard mpMRI confirmed on targeted or systematic biopsy
  Clinically significant prostate cancer is defined as Gleason Grade Group ≥ 2 (Gleason score ≥ 3+4 Predominantly well-formed glands with a lesser component of poorly-formed/fused/cribriform glands) based on histopathologic evaluation of biopsy cores obtained after PET/CT imaging.

SECONDARY OUTCOMES:
Incremental detection rate of csPCa by PET/CT over MRI | up to 6 months
  Proportion of participants in whom PET/CT leads to biopsy-confirmed csPCa (Grade Group ≥2) from a PET-positive / MRI-negative target measured by number of participants with csPCa detected on PET-positive, MRI-negative lesion from all participants who complete both imaging modalities and biopsy.
Lesion-level concordance between rhPSMA-7.3 (¹⁸F) PET/CT, multiparametric MRI, and histopathology | Up to 6 months following enrollment (from baseline imaging to confirmatory biopsy)
  Concordance (Yes/No) per lesion for location (lobe/zone/segment) and significance (csPCa yes/no on biopsy).
Predictive value of PET SUVmax for detecting clinically significant disease | Baseline to 6 months
  Comparing lesion-level concordance between PET/CT, mpMRI, and histopathology. Evaluating the predictive value of PET SUVmax for detecting clinically significant disease.
Sensitivity | Baseline to 6 months
  Sensitivity is defined as the probability of a positive PET/CT who actually have clinically significant disease.
Specificity | Baseline to 6 months
  Specificity is defined as the proportion of a true negatives on PET/CT who do not have clinically significant disease.
Positive Predictive Value (PPV) | Baseline to 6 months
  PPV is defined as the probability that a positive PET/CT is actually positive.
Negative Predictive Value (NPV) | Baseline to 6 months
  NPV is defined as the probability that a negative PET/CT is actually negative.
Number of participants that were reclassified | Baseline to 6 months
  Quantifying the proportion of patients reclassified (i.e., upgraded or transitioned from Active Surveillance (AS) to definitive treatment) based on PET/CT findings.

CONTACTS AND LOCATIONS:
Overall Officials: Ashutosh Tewari, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital / Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
The study involves a limited cohort of patients with localized prostate cancer undergoing advanced PSMA PET/CT imaging and confirmatory biopsy. Because the imaging and pathology data are inherently identifiable and linked to protected health information (PHI), sharing individual-level data could compromise participant confidentiality. Only aggregate, de-identified results will be shared through publications and presentations.